CLINICAL TRIAL: NCT00223782
Title: Motor Learning in Gait in Subjects With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Perell, Karen - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3117R
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Diabetes; Peripheral Neuropathy
Keywords: Diabetes; Peripheral Neuropathy; Walking
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases

ARMS (1):
- 1 (Other)
  Interventions: Behavioral: Gait Training with Feedback; Behavioral: Gait Training with no feedback

INTERVENTIONS:
Behavioral: Gait Training with Feedback
Behavioral: Gait Training with no feedback

SUMMARY:
The purpose of this study is to determine whether individuals with diabetic peripheral neuropathy can learn to change the way they walk in order to reduce the pressures underneath the feet, which may lead to a reduced risk of foot ulceration.

DETAILED DESCRIPTION:
This study suggests that teaching a new strategy is beneficial to decrease the forefoot peak plantar pressure in individuals who are susceptible to plantar ulcerations. It has not, however, been studied whether these changes would be maintained long-term or if they had any effect on the ulceration rate. Additionally, no analysis of the amount of visual feedback necessary to elicit the desired motor pattern was discussed. It has been suggested that proprioception plays an integral role in the use of feedback to develop error-detection mechanisms by integrating visual feedback and kinesthetic variables. In the diabetic peripheral neuropathy subject population, proprioception and kinesthesia may be compromised. This may have effects on the ability of this population to maintain changes in inappropriate movement patterns. A significant portion of patients continue to develop plantar ulcers even with prescriptive footwear compliance, so gait training to change inappropriate patterns which result in the high plantar pressures may be critical to prevent ulceration.

Comparisons: Two groups of subjects will receive gait training, one group will receive feedback of performance while the other will only receive training, and one control group. Comparisons will include whether plantar pressures are decreased in the training groups, and if those changes are maintained long-term.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diabetes for at least one year.
2. Diabetic peripheral neuropathy as defined by failure to sense the 5.07 (10g) monofilament test in one or more of the six sites tested (31;32)
3. Age 50-80 years old
4. Able to ambulate independently without assistive devices (e.g. walker or crutches) (8) for 30 feet.
5. No evidence of neurological (other than peripheral neuropathy) or orthopedic conditions

Exclusion Criteria:

1. Other non-diabetic causes of neuropathy by history
2. Symptomatic peripheral vascular disease
3. Joint pain, swelling and/or limited of range of motion in the lower extremities that interfere with walking or exercise
4. Visual problems not correctable with glasses or contact lens
5. Passive range of motion limitations are described as:

   1. Hip flexion < 1000;
   2. Hip extension < 200;
   3. Knee flexion < 1250;
   4. Knee extension < 00 (unable to obtain full extension);
   5. Ankle plantar flexion < 250;
   6. Ankle dorsiflexion < 150
6. Other systemic or local diseases that could interfere with walking assessment
7. Severe systemic diseases other than diabetes or its complications, especially those interfering with exercise tolerance
8. Amputation in the lower extremities
9. Terminal illness
10. Severe obesity: BMI>30 kg/m2 (33)
11. Severe foot deformities (e.g. flexion contracture of the toes, pes cavus, Charcot disease)
12. Mini-mental status of <27 or diagnosis of dementia
13. History of alcohol or drug abuse

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Plantar Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Karen Perell, PhD RKT, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States